CLINICAL TRIAL: NCT04591951
Title: A Family Navigator Intervention to Improve ADHD- Related Treatment Adherence (I2-ART) for Minority Children
Brief Title: Family Navigation to Improve ADHD Treatment Adherence for Minority Children
Acronym: I2-ART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Kelly Kamimura-Nishimura, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1K23MH125138-01 (NIH)
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Treatment adherence; Family navigation; Latinx; African American
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I2-ART Group (Active Comparator): I2-ART intervention will be modeled based on the Parent Empowerment Program model. It will use methods of adult learning, direct instruction to share knowledge or techniques for practice, group support, modeling, vicarious learning, and practice opportunities (i.e., role rehearsals). I2-ART training includes 40 hours of didactic and interactive sessions (10 sessions of 4 hours each) covering the following areas: 1) conceptual framework, 2) listening, engagement, and boundary-setting skills; 3) ADHD psychoeducation (e.g., diagnosis, treatment, shared decision-making tools), and 4) service options. The caregivers in the I2-ART group will receive the intervention for 3 months. The I2-ART will be implemented by the family navigators and will include a 2-hour face-to-face meeting, at least three monthly in-person meetings, and intermittent contact between in-person meetings by phone calls, texts or emails, as determined by the family navigator-caregiver dyad.
  Interventions: Behavioral: I2-ART
- Control Group (Placebo Comparator): The caregivers in the control group will receive "usual care."
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: I2-ART — Based on the Parent Empowerment Program model, I2-ART will use methods of adult learning, direct instruction to share knowledge or techniques for practice, modeling, vicarious learning, and practice opportunities (i.e., role rehearsals). The research team will provide the family navigators with 3 months of I2-ART training, including 40 hours of didactic and interactive sessions (10 sessions of 4 hours each). Following training, the family navigators will implement the 3-month I2-ART intervention with the caregivers, including a 2-hour face-to-face meeting, at least three monthly in-person meetings, and intermittent contact between in-person meetings by phone calls, texts or emails, as determined by the family navigator-caregiver dyad.
  Arms: I2-ART Group
Other: Usual care — Care as usual
  Arms: Control Group

SUMMARY:
ADHD is the most common pediatric neurodevelopmental disorder and is associated with significant long-term impairments. Current guidelines recommend stimulant medication and/or behavioral therapy as first-line treatments for ADHD. Despite evidence that consistent treatment is important for effectively managing ADHD symptoms, treatment adherence remains suboptimal and is especially problematic among minority children. Hypothesized reasons for racial/ethnic disparities in ADHD treatment include uncertainties about medication efficacy and side effects, distrust of the health care system, and decreased access to mental health services. This study aims to develop and test the I2-ART intervention to improve treatment adherence in minority (Latinx and African American) children with ADHD. The proposed study involves three ORBIT phases: During phase 1a, the investigators will conduct focus groups with key stakeholders (i.e., caregivers, clinicians, and family navigators, n=24) to identify and develop I2-ART's basic elements. Next, during phase 1b, the investigators will train four family navigators to implement I2-ART with caregivers of treatment-naïve children with ADHD (n=8-12) in order to determine feasibility and acceptability. In phase 2, the investigators will use phase 1b findings to modify I2-ART as needed, and then will evaluate the preliminary efficacy of the revised I2-ART (n=40), compared to the "usual care" control condition (n=20), on ADHD treatment adherence. The preliminary data collected during the proposed study will inform a subsequent R01 randomized controlled trial to examine I2-ART efficacy.

DETAILED DESCRIPTION:
The proposed project involves three phases consistent with the ORBIT model:

Phase 1a (9 months): The Parent Empowerment Program (PEP) developed by Dr. Hoagwood (consultant), has been tested in a diverse population of children and adults with mental illnesses, such as anxiety and depression, and has been shown to increase family empowerment, access to mental health services, and self-efficacy skills. However, PEP has not focused on ADHD care. The investigators will use the PEP program as I2-ART's foundation but specifically tailor the intervention to improve adherence to ADHD treatments using findings from the empirical literature regarding facilitators and barriers to adherence for African American (AA) and Latinx (Lx) youth with ADHD and their families. The investigators will gather feedback from the focus groups in Phase 1a to make adaptations to I2-ART and determine the most effective ways to deploy I2-ART, which will be needed to implement the intervention during Phase 1b. Focus groups participants (N=24) will include 6 clinicians (e.g., psychologists, general pediatricians, and developmental pediatricians), 6 experienced family navigators from prior PI and co-mentors' studies (3 Lx, 3 AA), 6 caregivers who are experienced with ADHD treatment for their child (3 Lx, 3 AA), and 6 caregivers of treatment-naïve children with ADHD (3 Lx, 3 AA). Eight focus groups will be conducted using the well-established Morgan & Krueger approach (e.g., group size of 3-6 participants). Separate focus groups will be conducted for each stakeholder group and for Spanish-speaking participants, including at least one focus group for clinicians, two for family navigators (1 Lx, 1 AA), and four for caregivers (2 Lx, 2 AA). First, the investigators will gather information from caregivers of children with ADHD who are experienced with ADHD treatment (Parent Focus Group 1) regarding their receptivity to collaboration with a family navigator as well as the most effective ways to introduce family navigator/caregiver dyads to each other and support their relationship. Then, the investigators will conduct focus groups with clinicians to obtain their perspective on needed PEP adaptations to address barriers to ADHD treatment adherence and how to identify patients within their clinical practices who may benefit from working with a family navigator. Next, the investigators will hold focus groups with family navigators to understand preferences for intervention delivery, including their feedback on the use of ADHD shared decision-making tools and animated videos to overview session key points with minority families. Feedback from all focus groups will be used to modify the I2-ART treatment manual and implementation plans, which will subsequently be reviewed by focus groups of caregivers of treatment-naïve children with ADHD (Parent Focus Group 2) for additional modifications. Throughout the focus groups, the investigators will use feedback to ensure I2-ART's cultural appropriateness. All focus groups will be facilitated by the PI and co-mentors experienced with focus groups (Drs. Modi, Crosby and Jacquez), and will last 1-2 hours. All sessions will be audio-/video-recorded, field notes composed, and sessions transcribed verbatim. The primary deliverable is the design and content for the I2-ART intervention, including a draft treatment manual.

Phase 1b (12 months): Four family navigators (2 Lx, 2 AA) will receive I2-ART training, and then will implement I2-ART with 2-3 culturally matched caregivers each (n=8-12). Feasibility, acceptability, and satisfaction with I2-ART will be assessed after intervention implementation. The investigators will make modifications to the I2-ART treatment manual based upon family navigator and caregiver feedback. Based on the PEP model, I2-ART will use methods of adult learning, direct instruction to share knowledge or techniques for practice, modeling, vicarious learning, and practice opportunities (i.e., role rehearsals). The research team will provide the family navigators with 3 months of I2-ART training, including 40 hours of didactic and interactive sessions (10 sessions of 4 hours each). The family navigators' I2-ART training will include these areas: 1) conceptual framework, 2) listening, engagement, and boundary-setting skills; 3) ADHD psychoeducation (e.g., diagnosis, treatment, shared decision-making tools), and 4) service options. Following training, the family navigators will implement the 3-month I2-ART intervention with the caregivers, including a 2-hour face-to-face meeting (session 1), at least three monthly in-person meetings (sessions 2, 3, and 4), and intermittent contact between in-person meetings by phone calls, texts or emails, as determined by the family navigator-caregiver dyad. Family navigators will meet weekly with research staff for supervision and case review. Family navigators and caregivers will complete questionnaires at baseline (B), after session 1 (Time 1), after session 2 (Time 2), after session 3 (Time 3), and immediately post-intervention (Time 4), and 3 months post-intervention (Time 5). In addition, the PI will interview the family navigators and caregivers to gain a more detailed understanding of their I2-ART experiences. After Phase 1b completion, the investigators will modify I2-ART as needed.

Phase 2 (24 months): Using a 2-wave approach, the investigators will evaluate the preliminary effectiveness of the revised I2-ART intervention, compared to a "usual care" control condition, on ADHD treatment adherence (e.g., initiation, implementation, and discontinuation of ADHD medication and/or behavioral treatment) in minority children (Lx, AA) with ADHD. Four family navigators (2 Lx, 2 AA) will implement the I2-ART treatment manual in 2 waves:

Wave 1 (12 months): Thirty caregivers (15 Lx, 15 AA) will be randomly assigned to the intervention group (n=20; 10Lx, 10AA) or "usual care" control group (n=10; 5Lx, 5AA). A research liaison at each recruitment site will request caregivers' permission for research staff to contact potential participants. Research staff will phone these families, and then meet face-to-face with those interested in study participation for informed consent. After enrollment, primary caregivers from both groups will meet with research staff to complete demographic and baseline measures (B). Then, for the intervention group, the family navigators will implement I2-ART for 3 months (including a 2-hour face-to-face meeting with the caregivers, at least three monthly in-person meetings, and intermittent contact between in-person meetings by phone calls, texts or emails). Family navigators will also meet weekly with research staff for supervision and case review. Caregivers in the control group will receive "usual care." In addition to completing the baseline surveys, family navigators and caregivers from both the intervention and control groups will complete questionnaires at Time 4 (immediately post-I2-ART for the intervention group) and Time 5 (3-months post-I2-ART for the intervention group).

Wave 2 (12 months): Thirty caregivers (15 Lx, 15 AA) will be randomly assigned to the intervention group (n=20; 10Lx, 10AA) or "usual care" control group (n=10; 5Lx, 5AA), and will use the same procedures as described for Wave 1.

Treatment fidelity will be measured through self-report from family navigators and caregivers, as well as through research staff assessment. For self-report, family navigators and caregivers will complete questionnaires to indicate whether they implemented/received identified intervention components. In addition, the investigators will audio record all family navigator/caregiver sessions (n=48 for Phase 1b, n=240 for Phase 2); then, the investigators will code 10% of the Phase 1b sessions (n=4) and 20% of the Phase 2 sessions (n=48) for fidelity. As with prior mentors' projects (Drs. Epstein and Froehlich),4,5 two independent coders (PI and research coordinator) will be trained and calibrated on the coding scheme and Noldus® software until reaching 90% reliability. The investigators will double code half of the coded sessions and will compute intraclass correlation coefficients to determine reliability of the fidelity coding. In addition, to ensure uniformity of intervention delivery, the investigators will develop an animated video using Vyond (an animated software tool) to provide an overview of core concepts and key points for each family navigator/caregiver session. This animated video overview of each session's contents will be viewed jointly by the family navigator and caregiver, and used as a springboard for discussion.

ELIGIBILITY:
1. Clinicians.

   Inclusion Criteria:
   * Currently providing care for children with ADHD as psychologists, general pediatricians, or developmental pediatricians.
   * > 18 years old.
   * Any race/ethnicity.

   Exclusion Criteria:

   * Unable to read/speak either English or Spanish.
2. Family navigators.

   Inclusion Criteria:
   * Having experience working as family navigator and/or community health worker.
   * Latinx (Lx) or African American (AA).
   * > 18 years old.

   Exclusion Criteria:

   * Unable to read/speak either English or Spanish.
3. Caregivers.

Inclusion Criteria:

* Phase 1a: current or former caregiver of a child with ADHD, with and without experience with ADHD treatment.
* Phases 1b and 2: current caregiver of a child (aged 7-11 years) with ADHD who is ADHD treatment-naïve at study enrollment.
* Lx or AA.
* > 18 years old.

Exclusion Criteria:

* Unable to read/speak either English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Intervention Sessions | 3 months after intervention, up to 6 months
  The family navigators will record the number of sessions attended by caregivers.
Length of Intervention Sessions | 3 months after intervention, up to 6 months
  The family navigators will record the length of sessions attended by caregivers.
Satisfaction with Intervention Immediately after Intervention | Immediately after intervention, up to 3 months
  This is a 7-item Likert scale questionnaire that elicits caregivers' and family navigators' opinions regarding the format, content, length, and convenience of the intervention. Answers ranged from Strongly Agree to Strongly Disagree. Higher score means better outcome (satisfaction).
Satisfaction with Intervention 3 months after Intervention | 3 months after intervention, up to 6 months
  This is a 7-item Likert scale questionnaire that elicits caregivers' and family navigators' opinions regarding the format, content, length, and convenience of the intervention. Answers ranged from Strongly Agree to Strongly Disagree. Higher score means better outcome (satisfaction).
System Usability Scale Immediately after Intervention | Immediately after intervention, up to 3 months
  The System Usability Scale is a 10-item Likert scale questionnaire that elicits family navigators' global views of the I2-ART treatment manual's usability. Answers ranged from Strongly Agree to Strongly Disagree. Higher score means better outcome (satisfaction).
System Usability Scale 3 months after Intervention | 3 months after intervention, up to 6 months
  The System Usability Scale is a 10-item Likert scale questionnaire that elicits family navigators' global views of the I2-ART treatment manual's usability. Answers ranged from Strongly Agree to Strongly Disagree. Higher score means better usability (outcome).
Family Navigator Activities Checklist | 3 months after intervention, up to 6 months
  This 27-item checklist will document family navigator-caregiver activities, including emotional support, action planning, information provision, advocacy, and skill development. Higher score means better outcomes (more activities covered by family navigators).
Implementation Questionnaire | 3 months after intervention, up to 6 months
  The implementation questionnaire will include 10 items recording information about treatment fidelity, time needed for the intervention, enrollment rate, reasons for declining participation, representativeness of the sample, facilitators/barriers to delivering the I2-ART intervention, facilitators/barriers for sustaining intervention after study completion, feedback regarding intervention. Higher score means better implementation (outcome).
Change in Services Use in Children and Adolescents from Immediately after Intervention to 3 months after Intervention | Immediately after intervention (up to 3 months) and 3 months after intervention (up to 6 months)
  This structured interview assesses use of services for mental health and related issues (e.g., medication and/or behavior therapy).
ADHD medication initiation immediately after intervention | Immediately after intervention, up to 3 months
  We will obtain data regarding ADHD medication initiation based on Prescription Drug Monitoring Program records and medical chart review.
ADHD medication initiation 3 months after intervention | 3 months after intervention, up to 6 months
  We will obtain data regarding ADHD medication initiation based on Prescription Drug Monitoring Program records and medical chart review.
Percent of days covered with ADHD medication immediately after intervention | Immediately after intervention, up to 3 months
  We will obtain data regarding percent of days covered with medication once initiated based on Prescription Drug Monitoring Program records.
Percent of days covered with ADHD medication 3 months after intervention | 3 months after intervention, up to 6 months
  We will obtain data regarding percent of days covered with medication once initiated based on Prescription Drug Monitoring Program records.
Discontinuation of ADHD medication immediately after intervention | Immediately after intervention, up to 3 months
  We will obtain data regarding discontinuation of medication once initiated based on Prescription Drug Monitoring Program records and medical chart review.
Discontinuation of ADHD medication 3 months after intervention | 3 months after intervention, up to 6 months
  We will obtain data regarding discontinuation of medication once initiated based on Prescription Drug Monitoring Program records and medical chart review.
Behavior Therapy Initiation immediately after intervention | Immediately after intervention, up to 3 months
  Through medical chart review, we will obtain data regarding initiation of behavior therapy when recommended by clinician.
Behavior Therapy Initiation 3 months after intervention | 3 months after intervention, up to 6 months
  Through medical chart review, we will obtain data regarding initiation of behavior therapy when recommended by clinician.
Number of Behavior Therapy Visits immediately after intervention | Immediately after intervention, up to 3 months
  We will obtain data regarding the number of behavior therapy visits attended by family through medical chart review.
Number of Behavior Therapy Visits 3 months after intervention | 3 months after intervention, up to 6 months
  We will obtain data regarding the number of behavior therapy visits attended by family through medical chart review.
Behavior Therapy Disengagement immediately after intervention | Immediately after intervention, up to 3 months
  We will obtain data regarding behavior therapy disengagement through medical chart review.
Behavior Therapy Disengagement 3 months after intervention | 3 months after intervention, up to 6 months
  We will obtain data regarding behavior therapy disengagement through medical chart review.

SECONDARY OUTCOMES:
Change in Vanderbilt ADHD Parent Report Scale Scores from baseline to 3 months after intervention | Baseline and 3 months after intervention
  The Vanderbilt ADHD Parent Report Scale is a 25-item scale that assess ADHD symptoms, including 9 attention items and 9 hyperactivity/impulsive items. Answers ranged from (0) Never to (3) Very Often. Summary scores for the 2 ADHD symptom domains are created by summing the 9 inattention and the 9 hyperactivity/impulsivity items.

OTHER OUTCOMES:
Working Alliance Inventory | Baseline, after first session (up to 1 week), after intervention session (up to 1 month), after third session (up to 2 months), immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  The Working Alliance Inventory is a 12-item measure of a family's perceived agreement with their healthcare provider on the goals/tasks of treatment and the extent to which they have a strong personal bond with their provider. Respondents rate their responses on a scale of 1 (strongly disagree) to 5 (strongly agree). Item scores are summed, giving a range from 12-60, with higher scores indicating a better family-provider alliance.
Family Empowerment Scale | Baseline, after first session (up to 1 week), after intervention session (up to 1 month), after third session (up to 2 months), immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  The Family Empowerment Scale is a 12-item scale that assess perceptions and attitudes about family navigator and caregiver roles/responsibilities within their local service systems and their ability to advocate on behalf of their children. Items are scored on a 5-point likert type scale from 1 (Never) to 5 (Very often). The FES assesses three domains, Work (e.g. "I know what to do when problems arise with the families with whom I work"), Children's Services (e.g., "I make sure that professionals understand caregivers' opinions about what services their children need"), and Community (e.g. "I feel I can have a part in improving services for children in my community").
Collaborative Skills Questionnaire | Baseline, immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  The Collaborative Skills Questionnaire is a 36-item scale examining key knowledge and skills development related to training modules. It includes six subscales, one for each I2-ART training manual module: (1) Listening, Engagement, and Boundary Settings Skills, (2) Group Management, (3) Priority Setting, (4) Specific Disorders and Their Treatment, (5) Mental Health Services, and (6) School Options. Questions include, "I can talk to parents about our mutual responsibilities in the working relationship" and "I am aware of barriers that parents may face in seeking help for their children and know how to help them overcome those barriers."
Vanderbilt Mental Health Services Efficacy | Baseline, immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  This 25-item scale examines the degree to which family navigators and caregivers feel effective in accessing mental health services. Items are scored on a five-point scale from 1 (strongly disagree) to 5 (strongly agree). Typical items include, "I believe that I can help parents access and use effectively mental health services for their children" and "My skills in dealing with mental health services will help me to empower parents to change things that might be wrong with their child's treatment."
Brief Illness Perceptions Questionnaire | Baseline, after first session (up to 1 week), after intervention session (up to 1 month), after third session (up to 2 months), immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  This 11-item scale is designed to assess a parent's representation of ADHD (e.g. expected time course, consequences, causes, etc.). It has good test-retest reliability as well as concurrent and predictive validity. All of the items, except the causal scale, are rated using a 0 to 10 response scale. For the causal scale, parents list the three most important causal factors in their child's ADHD/ADD, and responses are grouped into categories (genetic, environmental, behavioral, dietary, etc.) for analysis.
Beliefs about Medicines Questionnaire | Baseline, immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  The validated 25-item Beliefs about Medicines Questionnaire has two domains, Specific and General. The BMQ-Specific comprises two scales: 1) Necessity (parent beliefs about the necessity of prescribed medication) and 2) Concerns (parent concerns about potential adverse consequences of using medication). The BMQ-General comprises two scales: 1) Overuse (parent beliefs about overuse of medicine by doctors) and 2) Harm (parent belief about the intrinsic harmfulness of medicine). For all items on all scales, respondents indicate their degree of agreement with each individual statement on a 5-point Likert-type scale (e.g., 1=strongly disagree to 5=strongly agree). Scores obtained for the individual items within each scale are summed to give a scale score. Mean scores are also calculated for each scale (range of 1 to 5). In addition, a Necessity/Concerns Differential (NCD) is calculated by subtracting the mean Concerns scale score from the mean Necessity scale score (range of -4 to 4).
Decisional Conflict Scale | Baseline, immediately after intervention (up to 3 months), 3 months after intervention (up to 6 months)
  This 16-item validated measure elicits the parent's preference for treatment options and parent-perceived sources of decisional conflict about their preferred option. The scale produces a total score with five subscales: 1) informed; 2) values clarity; 3) support; 4) uncertainty; 5) effective decision. Lower scores are desirable, with a range from 0-100.
Participants' Age | Baseline
  Through the Background History Form, the investigators will collect the family navigators' and caregivers' age.
Participants' Race and Ethnicity | Baseline
  The Background History Form will collect family navigators' and caregivers' race and ethnicity.
Participants' Employment Status | Baseline
  The Background History Form will collect family navigators' and caregivers' employment status.
Caregivers' Income | Baseline
  The Background History Form will collect caregivers' household income.
Caregivers' Educational Level | Baseline
  The Background History Form will collect caregivers' educational level.
Caregivers' Marital Status | Baseline
  The Background History Form will collect caregivers' marital status.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Kamimura-Nishimura, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No